CLINICAL TRIAL: NCT04747028
Title: Effect of Malnutrition on Primary and Permanent Dentition a Cross Sectional Study
Brief Title: Effect of Malnutrition on Primary and Permanent Dentation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina mounir elkady, Lecturer at conservative department, Cairo University
Other Study IDs: 66789
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Study Focus on the Effect of Malnutrition and Dental Problem

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Primary dentition: Children from 4 to 6 years old suffering from malnutrition
  Interventions: Diagnostic Test: Dmf score
- Age 13 to 16: Adolecentsfrom 13 to 16 suffering from malnutrition at present time or during their childhood
  Interventions: Diagnostic Test: Dmf score

INTERVENTIONS:
Diagnostic Test: Dmf score — A chart to calculate the caries index

SUMMARY:
The caries index delayed eruption and enamel malformation will recorded for a 2 group of participants

DETAILED DESCRIPTION:
The participants suffering from malnutrition will be divided into age group from 4 to 6 to study the primary dentition and another group age from 13 to 16to study the primary dentition caries index with dmf and DMF score Modified DDE index for measurement of developmental defects in enamel

ELIGIBILITY:
Inclusion Criteria:

* parent accept to sign the informed consent Participants not suffering from any other systematic disease

Exclusion Criteria:

* non coopreative patient Suffering from systematic disease

Ages: 4 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Children and adolescent diagnosed with malnutrition in the past or presnt time.patient should not suffer from any other systemic disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Caries index | 1month
  Score obtained from DMF index

SECONDARY OUTCOMES:
E amel malformation | 1month
  Modified DDE index

IPD SHARING:
Plan to Share IPD: Undecided